CLINICAL TRIAL: NCT03907059
Title: Does Exclusive Consumption of Plant-based Dietary Protein Impair Resistance Training-induced Muscle Adaptations?
Brief Title: Plant-based Dietary Protein and Resistance-training Adaptations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 54014116.9.0000.5391
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Healthy
Keywords: protein source; hypertrophy; resistance training; plant-based protein; omnivorous
MeSH Terms: conditions — Hypertrophy | interventions — Whey Proteins; Soybean Proteins

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omnivorous (Active Comparator): Interventions: Daily protein intake was adjusted to 1.6g/kg/day via supplementation (whey) + 12 weeks of resistance training
  Interventions: Dietary Supplement: whey protein
- Vegan (Experimental): Interventions: Daily protein intake was adjusted to 1.6g/kg/day via supplementation (soy) + 12 weeks of resistance training
  Interventions: Dietary Supplement: soy protein

INTERVENTIONS:
Dietary Supplement: whey protein — supplementation individually adjusted to 1.6g/kg/day
  Arms: Omnivorous
Dietary Supplement: soy protein — supplementation individually adjusted to 1.6g/kg/day
  Arms: Vegan

SUMMARY:
Dietary protein consumption maximizes the anabolic response during resistance training (RT) by triggering muscle protein synthesis and providing the indispensable amino acids for a net positive protein balance. Leucine is considered the key amino acid in this process, suggesting that differences in protein quality may influence RT-induced gains in muscle mass and strength. In general, plant-based protein sources have lower leucine concentrations than animal-based protein sources and human skeletal muscle. In this respect, despite acute evidence on lower anabolic properties of plant- vs. animal-based protein, the effects of an exclusive plant-based dietary protein diet on RT-induced adaptations are currently unknown.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young men
* Vegans ≥ 1 y or omnivorous subjects
* Physically active but no resistance-trained subjects
* Without any chronic injury that impairs resistance training performance
* Protein intake > 0.8 g/protein/kg body weight

Exclusion Criteria:

* Use of creatine or beta-alanine supplements for the last 3 months
* Use of proteins and/or amino acids supplements for the last 1 month
* Engagement in specific dietary restrictions
* Previous use of anabolic steroids
* Engagement in any training program

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Muscle cross-sectional area | 12 weeks
  assessed by mode-B ultrasound
Muscle strength | 12 weeks
  assessed by leg-press one-maximum-repetition

SECONDARY OUTCOMES:
Leg lean mass | 12 weeks
  assessed by Dual-energy X-ray absorptiometry
fiber cross-sectional area | 12 weeks
  assessed by muscle biopsy (vastus lateralis)

CONTACTS AND LOCATIONS:
Overall Officials: Hamilton Roschel, Professor, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Hevia-Larrain V, Gualano B, Longobardi I, Gil S, Fernandes AL, Costa LAR, Pereira RMR, Artioli GG, Phillips SM, Roschel H. High-Protein Plant-Based Diet Versus a Protein-Matched Omnivorous Diet to Support Resistance Training Adaptations: A Comparison Between Habitual Vegans and Omnivores. Sports Med. 2021 Jun;51(6):1317-1330. doi: 10.1007/s40279-021-01434-9. Epub 2021 Feb 18. PMID 33599941